CLINICAL TRIAL: NCT00294424
Title: A Prospective, Multi-Centre Study on Costs and Effects of Waiting Time in Patients Undergoing Total Hip and Knee Replacement Surgery. A Randomized Controlled Trial.
Brief Title: Study on Costs and Effects of Waiting Time in Total Hip and Knee Replacements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academy of Finland (Other)
Collaborators: Hospital District of Helsinki and Uusimaa (Other); Coxa, Hospital for Joint Replacement (Other); Tampere University (Other); Orton Invalid Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AF51871
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2006-01

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis, Knee
Keywords: Waiting time; Total hip replacement; Total knee replacement; Quality of life; The15D; Harris Hip Score; Knee Score; Pain measurement; Cost-effectiveness; Medication; Health services; Social services; Randomized Controlled Trial
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

INTERVENTIONS:
Procedure: Short waiting time
Procedure: Non-fixed waiting time

SUMMARY:
The aim of this study is to compare the cost-effectiveness of major joint replacement in patients with short and non-fixed (control group) waiting time (WT). After being placed on the waiting list, patients will be randomized into two groups through regular contact with the practice staff: (1) Patients with non-fixed waiting time (patient undergoes hospital's normal procedure from the date (s)he is added to the waiting list to the date of operation), and (2) patients with short waiting time (operated in maximum three months). The main question is: is it possible to improve the cost-effectiveness of major joint replacement by shortening waiting time?

DETAILED DESCRIPTION:
The aim of this study is to compare the cost-effectiveness of major joint replacement in patients with short and non-fixed (control group) waiting time (WT). After being placed on the waiting list, patients will be randomized into two groups through regular contact with the practice staff:

1. Patients with non-fixed waiting time (patient undergoes hospital's normal procedure from the date (s)he is added to the waiting list to the date of operation), and
2. patients with short waiting time (operated in maximum three months).

For ethical reasons, care will be taken to avoid any risk of inequality between the patient groups. Such inequality might result if some patients should wait for access to treatment longer than normally or if short waiting times would accounted for more than half of the hospital's surgical capacity, for instance. The number of patients placed on the waiting list varies from one month to another, being specific to each hospital. Therefore no advance estimate can be made of the number of patients to be placed on the list. Consequently, the following arrangements will be made:

1. the patients randomised into the short WT group could only be operated on every fourth month, and only half of the hospital's one-month surgical capacity could be allocated as short WTs, so the number of short WTs will be restricted and determined specifically for each hospital;
2. it will be ensured that all eligible patients placed on the waiting list have a chance of getting recruited into the study (including the possibility of short WT) by not restricting the size of the non-fixed WT group. In order to avoid selection bias among the patients, the groups will be different in size.
3. Recruitments will be made in periods of three months in order to avoid the waiting time for the short WT group exceeding three months.

Randomization is made by the nurse responsible using consecutively numbered and sealed envelopes. Participants complete a self-administered questionnaire at four specific points in time:

1. when placed on the waiting list by the orthopaedic surgeon (baseline),
2. at hospital admission,
3. three, and
4. 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* a need for a primary unilateral or bilateral THR (total hip replacement) or TKR (total knee replacement) due to osteoarthritis (OA) evaluated by the orthopaedic surgeon
* aged 16 years or older
* female or male
* patient is placed on the waiting list in a research hospital
* the patent is willing and mentally able to participate in the study.

Exclusion Criteria:

* Subjects with rheumatoid arthritis
* Subjects with fractures
* Subjects with haemophilia
* Subjects with congenital deformities
* Subjects with a need for re-arthroplasty

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 833
Dates: Start 2002-09; Study Completion 2006-04

PRIMARY OUTCOMES:
The generic, 15-dimensional and standardised health status instrument 15D
when placed on the waiting list, at admission, 3 months and 12 months after surgery

SECONDARY OUTCOMES:
Modified Harris Hip Score
Modified Knee Score
10-cm horizontal visual analog scale (VAS)
Perceived health on a scale 1-5: excellent, very good, good, moderate and poor
Use and costs of health services
Use and costs of social services
Use and costs of informal care
Use and costs of medication
Patients' demographic characteristics like:
-age
-gender
-education
-marital status
-employment status
-BMI (body mass index)
-co-morbidity
-housing
-home municipality
when placed on the waiting list, at admission, 3 months and 12 months after surgery
Hospital costs during hospital treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marja L Blom, PhD, Study Director — Academy Of Finland/ Stakes/ National Research and Development Centre for Welfare and Health
Locations (1):
- Stakes/National Research and Development Centre for Welfare and Health, Helsinki, Helsinki, Finland

REFERENCES:
- [Background] Sintonen H. 2001. The 15D instrument of health-related quality of life: properties and applications. The Finnish Medical Society Duodecim, Ann Med 33: 328-336 Sintonen H. http://www.15d-instrument.net/15d Drummond M. 2001. Introducing economic and quality of life measurements into clinical studies. Ann Med 33: 344-353 Mahomed NN, Arndt DC, McGrory BJ, Harris WH. The Harris Hip Score. Comparison of patient self-report with surgeon assessment. J Arthroplasty 2001; 16: 575-580 Insall JN, Lawrence DD, Scott RD, Scott WN. 1989. Rationale of The Knee Society Clinical Rating System. Clin Orthop. 248: 13-14 McDowell I, Newell C. 1996. Measuring Health: A Guide to Rating Scales and Questionnaires, 2nd edn. New York: Oxford University Press Hujanen T. Unit cost of health care in Finland 2001. Helsinki: Stakes. Aiheita 1/2003 (in Finnish) Pharmaca Fennica. CD-Pharmaca. 2004. Lääketietokeskus (in Finnish)